CLINICAL TRIAL: NCT06712966
Title: EngageRx With Integrated Self-Measurement of Blood Pressure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study deemed not human subjects research and will proceed as quality improvement.
Sponsor: University of California, San Francisco (Other)
Collaborators: New York University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-42835; 1R43DP006817-01 (NIH)
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-04-07 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Single-arm interventional study with comparison to historical controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EngageRx_SMBP (Experimental): Integrated SMBP monitoring using EngageRx_SMBP.
  Interventions: Other: EngageRx_SMBP

INTERVENTIONS:
Other: EngageRx_SMBP — Patients in the EngageRx_SMBP arm will be automatically registered in the CareSimple system and mailed a device they can use at home. They may also choose to install a smartphone application from CareSimple that will provide reminders about measuring their BP. The clinician will then manage the patient's hypertension according to the standard of care. The SMBP measurements from CareSimple will be available through EngageRx for them to use, and they will receive a weekly staff message to check EngageRx if there are new SMBP measurements for them to review. The clinician will also be able to indicate when they would like to stop using the CareSimple system.

SUMMARY:
This pilot study will support use of EngageRx_SMBP for 70 patients in the UCSF General Internal Medicine practice. The goals of the pilot will be to assess usability and satisfaction of both patients and clinicians, and to describe BP-related process metrics and outcomes including time to intensification of BP medications and/or BP control.

DETAILED DESCRIPTION:
EngageRx is a programmable clinical decision support app that clinicians can access within the context of their electronic health record (EHR), and it can be connected with other technologies. We are integrating EngageRx with CareSimple, a company that provides a cellular-enabled BP device that patients can use for SMBP. CareSimple devices are FDA-cleared, can be shipped directly to patients, used by patients right out of the box (after installing batteries), and then deliver the SMBP measurements directly to the CareSimple cloud platform. There is no requirement to "sync" the device, and no need for patients to have a smartphone or set up an account or sign into anything. CareSimple supports a dashboard and portal that allows authorized users to sign in and access measurements for a patient, but this amounts to another barrier for clinicians to access the measurements; our integration with EngageRx will 1) allow clinicians to initiate SMBP monitoring for a patient with the click of a button (after confirming their shipping address and preferred language); 2) automatically register the patient in the CareSimple system, which triggers CareSimple to mail the patient the BP monitor device with instructions; and 3) automatically push the CareSimple SMBP measurements to EngageRx so they are available the next time the clinician opens EngageRx. The SMBP measurements will be used with EngageRx's internal algorithm, along with office BP measurements, to recommend BP management decisions to clinicians. We believe this integrated system, which we will refer to as EngageRx_SMBP, will make SMBP easy for clinicians and patients. We would like to determine if this system is truly easy to use for clinicians and providers, and whether it appears to facilitate the BP-related processes of care required for controlling hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18+ years old) with uncontrolled BP in an office visit
* Lowest SBP>140 or lowest DBP>90 during the visit at one of the Mt. Zion General Internal Medicine practices
* Speaks English or Spanish

Exclusion Criteria:

* If patient is unlikely to be able to use a home BP monitor
* Cannot understand the verbal consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Net Promoter Score | 3 months
  This score is assessed by asking a single question about likelihood of recommending the device to a friend, with options from 1-10 (10 being extremely likely). As per published methods, persons indicating 9 or 10 are considered "Promoters"; persons indicating 7 or 8 are "Passives"; and persons indicating 1-6 are "Detractors". The score is calculated by taking the percent of Promoters and subtracting the percent of Detractors, yielding a score for each group ranging from -100 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pletcher, MD MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamilton DF, Lane JV, Gaston P, Patton JT, Macdonald DJ, Simpson AH, Howie CR. Assessing treatment outcomes using a single question: the net promoter score. Bone Joint J. 2014 May;96-B(5):622-8. doi: 10.1302/0301-620X.96B5.32434. PMID 24788496
- [Background] Krol MW, de Boer D, Delnoij DM, Rademakers JJ. The Net Promoter Score--an asset to patient experience surveys? Health Expect. 2015 Dec;18(6):3099-109. doi: 10.1111/hex.12297. Epub 2014 Oct 27. PMID 25345554